CLINICAL TRIAL: NCT03816150
Title: Interventions to Reduce Sedentary Behavior at Work: Pilot Study
Brief Title: Reduce Sedentary Behavior at Work
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jacquelyn Kulinski, Associate Professor, Medical College of Wisconsin
Other Study IDs: 25912
Record Dates: First submitted 2019-01-17; First posted 2019-01-25 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Sedentary Lifestyle; Obesity; Cardiovascular Risk Factor
MeSH Terms: conditions — Sedentary Behavior; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood (10 ml) and urine (10cc)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prior research suggests that sedentary behavior is detrimental to health, independent of exercise activity. Sedentary behavior is defined as behaviors that involve low levels of energy expenditure ≤1.5 metabolic equivalents (including sitting, watching TV, reading, and driving). Due to the high burden of sedentary behaviors in modern-day societies, this has potential implications for novel intervention strategies to reduce sitting (outside of regular exercise activity) and improve health. In addition, the modern workplace fosters sedentary behavior, and sedentary jobs now make up more than 80% of the workforce. The goal of this project is to implement interventions to reduce sedentary behavior at work and evaluate their impact on physiologic parameters and markers of disease. Specifically, the investigators/study team will use direct measurement of vascular endothelial function as one of our outcomes. This is important since conduit artery endothelial function, assessed by arterial flow-mediated dilation (FMD), is a powerful indicator of vascular inflammation and predictor of future cardiovascular events.

DETAILED DESCRIPTION:
The hypothesis is that obese subjects with sedentary jobs at the Medical College of Wisconsin, when assigned use of a standing desk to encourage movement, will reduce their daily sedentary time and demonstrate improvement in physiologic parameters and disease markers from baseline through the end of the intervention.

Prior intervention studies are limited and not randomized, but have shown a reduction in waist circumference and improvements in cholesterol when overall sitting time is reduced over a 3-6 month interval (with a standing or treadmill desk). None of these intervention studies have directly measured vascular endothelial function, as assessed by arterial flow-mediated dilation (FMD), an early indicator of cardiovascular disease, and a powerful predictor of future cardiovascular events and vascular inflammation. Improvements in arterial FMD (or endothelial function) are known to reduce the future risk of cardiovascular events.

Due to differences in the energy requirement of lying down, sitting, and standing, there has been increased research interest in activity type classification based on posture. In the science of sedentary behaviors, this is an important distinction to consider when evaluating health outcomes, such as in the present study. Accelerometers (physical activity monitors) utilize piezoelectric crystal sensor technology to provide a measure of accelerations of the body during movement and have the advantage of capturing frequency, duration, and intensity of physical movement minute by minute. Accelerometer technology will be used to analyze the primary outcome of interest (sedentary time). The study team will collect information on standing time, sedentary bouts, daily steps, cadence (walking speed in steps/minute), and exercise activity. The study team will employ a compact and re-usable physical activity monitor that adheres to the subject's thigh. This will provide objective assessments of activity levels at baseline and during the intervention. This data can be translated into energy expenditure or activity intensity categories (METs) and even position (sitting verses standing). The monitor output is Excel-compatible and is ideal for comparing each subject's activity and physiological parameters from baseline to intervention.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary office workers the Medical College of Wisconsin who spend greater than 75% of their (8 hours or longer) work-day sitting at a desk. This includes at least 1 period of 2 hours or longer of uninterrupted sitting time per work day.
* Body mass index of 26.0-44.9
* Willing and able to sign Informed consent
* Permission from the subject's supervisor to participate in the intervention

Exclusion Criteria:

* Known history of atherosclerotic cardiovascular disease, including myocardial infarction, stroke, coronary stent, coronary artery bypass grafting, angina and peripheral vascular disease
* Diabetics on insulin or other diabetic medications (pre-diabetes would be acceptable, defined as a HbgA1c of 5.7 to 6.4%, and not on medications)
* Elevated blood pressure (SBP≥150 mm Hg or DBP ≥90 mm Hg) or on medication for hypertension; or SBP < 100 mm Hg.
* On cholesterol-lowering medication or LDL-C cholesterol ≥190 mg/dL
* Pregnancy, lactating or planning to get pregnant within the next 6 months
* Current tobacco use within previous 12 months. Tobacco use included cigarettes, cigars, and all forms of smokeless tobacco.
* Current excessive alcohol use (defined as more than 14 drinks/week for women, more than 28 drinks/week for men)
* Current illicit drug use, defined as overuse of prescription medications, or of any illegal mind altering substances.
* Known thyroid disease
* Taking diet pills, or supplements other than those contained in a multi-vitamin
* History of musculoskeletal surgery/injury that would interfere with prolonged periods of standing
* History of use of PDE-5 inhibitors for any reason within the last 5 days of screening visit, and the inability to hold use of PDE-5 inhibitors for 5 days prior to each of the FMD evaluations.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sedentary office workers at the Medical College of Wisconsin who spend greater than 75% of their (8 hours or longer) work-day sitting at a desk.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
The feasibility of implementing workplace interventions to reduce sedentary time, specifically using a sit-stand desk. We will survey the subjects regarding the feasibility and likability of the sit-stand workstation | through study completion, an average of 6 months
  Ten Questions using a Likert Scale. Each question has the same 5 options: strongly agree, agree, neutral, disagree, strongly disagree.
The feasibility of implementing workplace interventions to reduce sedentary time, specifically using a sit-stand desk. We will survey the subjects regarding the feasibility and likability of the sit-stand workstation | Change from baseline sedentary behaviors after 6 months
  Objectively quantify sitting, standing and walking times (sedentary vs. non-sedentary) using an accelerometer device that adheres to the subjects thigh

SECONDARY OUTCOMES:
The Impact of reducing sedentary time on physiological outcomes | Change from baseline after use of a standing desk, through study completion, an average of 6 months
  Measure Flow Mediated Dilation (FMD)
The Impact of reducing sedentary time on physiological outcomes | Change from baseline after use of a standing desk, through study completion, an average of 6 months
  Measure Near-infrared spectroscopy is a spectroscopic (NIRS)
The Impact of reducing sedentary time on physiological outcomes | Through study completion, an average of 6 months
  anthropometrics: Change from baseline body mass index after use of a standing desk
The Impact of reducing sedentary time on physiological outcomes | Through study completion, an average of 6 months
  measure cardiac hemodynamics: Change from baseline systolic and diastolic blood pressure after use of a standing desk,
The Impact of reducing sedentary time on physiological outcomes | Through study completion, an average of 6 months
  measure cardiac hemodynamics: Change from heart rate after use of a standing desk,
The Impact of reducing sedentary time on physiological outcomes | At baseline after use of a standing desk, through study completion, an average of 6 months
  Measure blood lab results: Change from baseline fasting lipids, insulin resistance, hemoglobin A1c and C-reactive protein (CRP)